CLINICAL TRIAL: NCT03953534
Title: Quantity of Opioids for Acute Pain and Limit Unused Medication (OPUM Study)
Brief Title: Quantity of Opioids for Acute Pain and Limit Unused Medication
Acronym: OPUM
Status: Completed | Type: Observational
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Queen's University (Other); Maisonneuve-Rosemont Hospital (Other); Sunnybrook Health Sciences Centre (Other); Hopital de l'Enfant-Jesus (Other)
Responsible Party: Principal Investigator, Raoul Daoust, Clinician Researcher, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Other Study IDs: 2019-1684; PJT-159808 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2019-05-10; First posted 2019-05-16 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Acute Pain
Keywords: Opioids; Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Opioids (morphine and morphine-like substances) are often prescribed to patients to manage pain after an emergency department visit. In the past 20 years, opioid prescriptions have risen sharply, accompanied by a significant rise in opioid misuse (e.g., recreational or non-medical use, potentially leading to addiction or overdose). One explanation for this crisis is the availability and easy access of leftover opioid pills in Canadian homes, allowing family members (including children) and friends to take them for reasons other than pain relief.

Canada has no recommendations for the dosage, duration, or quantity of opioids that physicians should prescribe to manage acute pain at home. Physicians are therefore left guessing as to how much to prescribe when a patient with a condition like a fracture or renal colic is discharged from the emergency department. Our preliminary study showed that two-thirds of the pills from the initial opioid prescription to treat acute pain actually remained unused and were therefore available for potential misuse.

The investigators propose to determine how many opioid pills are consumed by patients who suffer from acute pain as they recover at home. The investigators will ask 2,560 patients (from 6 Canadian hospitals) to record their pain medication consumption in a 14-day diary. The investigators will also determine, their pain intensity level, whether or not they had new opioid prescriptions, and health services revisits. In case of missing information, patients will be contacted by phone at 2 weeks. The overall aim is to help emergency department physicians prescribe the right number of pills in order to manage patients' pain and at the same time reduce substantially leftovers available for potential misuse.

DETAILED DESCRIPTION:
Introduction

Prescription opioid overdoses have quadrupled in the last 15 years, and are now the leading cause of accidental death, surpassing motor vehicle accidents. The drastic rise in opioid prescription rates in Canada and the US could be the driving force behind this higher mortality. It was shown that 71% of opioid misusers (i.e., intentional users for nonmedical purposes) received their drugs through the diversion of unused prescribed opioids (transfer of opioids to someone other than the holder of the initial prescription). Emergency department (ED) physicians are among the top opioid prescribers for patients under 40, and there are currently no prospective studies on how many opioid pills should be prescribed to patients discharged from the ED with common pain conditions in order to limit unused pills. Preliminary results from our group revealed that two-thirds of the total prescribed opioids were not consumed and remained available for misuse.

Objectives

The ultimate goal of this research program is to decrease opioid misuse by lowering the quantity of unused medications. The primary objective of this project is to determine the quantity of opioids consumed during the acute pain phase (2 weeks) by ED-discharged patients treated for an acute pain condition. The secondary objectives are to inventory the quantity of opioids prescribed and unused after ED visits, use of co-analgesics, pain intensity, health services revisits during the 2-week follow-up, and chronic pain prevalence at 3 months.

Methods

The investigators propose a multicentre prospective observational cohort study in 2,560 consecutive ED patients recruited from 6 Canadian hospitals. The study will include patients aged ≥18 years, treated for an acute pain condition present for less than 2 weeks (usual acute pain definition), and discharged from the ED with an opioid prescription. Pain at triage and at ED discharged, diagnosis, and complete pain medication prescription will be initially listed. Patients will complete a 14-day electronic diary using the REDCap web-based system to document their daily pain medication consumption, pain intensity, new opioid prescriptions, and health services revisits. Patients will also answer questionnaires at 2 weeks and 3 months for our various secondary objectives. To validate the patient self-report opioid consumption, a randomized subset of patients will come back to the emergency for a follow-up visit and a manual count of the remaining opioids. As mitigation strategies (validated in our pilot study), non-responders to the diary will be contacted by phone at 2 weeks to answered questions summing diary information, and paper versions will be available for patients without Internet access.

Sample size estimation

The sample size was calculated to obtain an accurate estimate of the mean quantity of 5 mg morphine pill equivalent that patients will consume during the first 2 weeks after ED visit for each pain condition (primary objective). Our preliminary study was used to determine the standard deviation of opioids consumed after discharge from ED (SD=16). To estimate the mean 5 mg morphine pill equivalent consumed for each of the five pain conditions (acute back pain, fracture, sprain/contusion, renal colic, and other) with a 95%CI margin of error of 1.5 pills (or ~10% of the SD) with a standard deviation of 16 pills, each diagnostic category requires 440 patients. With the 14% attrition rate observed during our pilot study at two weeks, a total of 2,560 patients will be recruited (512 patients - 72 lost to follow-up = 440 patients per pain condition). Sample size calculations were performed using PASS (Power Analysis & Sample Size software, version 11.0: NCSS Statistical Software).

Feasibility

The investigators demonstrated the study feasibility in a successful pilot study with 627 patients at our academic ED. Additionally, our project brings together a committed, multidisciplinary research team, and all proposed study sites have collaborated previously on large multicentre studies. Finally, all instruments have been successfully tested, allowing rapid study implementation.

Impact

Our results will determine the quantity of opioids consumed during the acute pain phase (2 weeks) to ED-discharged patients treated for acute pain conditions. Our team members from relevant provincial and national stakeholders and patient associations, our strong evidence, and our extensive knowledge transfer strategy have the potential to impact physicians' opioid prescription practices. Consequently, fewer unused prescription opioids should lead to a substantial decrease in the currently high rate of opioid misuse.

ELIGIBILITY:
Inclusion Criteria:

* Opioid prescription at discharge
* Acute pain for less than 2 weeks

Exclusion Criteria:

* Language barrier
* Chronic pain under treatment
* Active Neoplasia
* Follow-up impossible / Unable to complete agenda
* Already on opioids

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — The patient's sex/gender may have an incidence on the quantity of opioids consumed. We will also look if there are sex/gender differences in the quantity of opioids prescribed and unused, in pain trajectory, in reasons for stopping opioids, and access to the health care system.
  The patient gender will be self-reported in the electronic diary (or paper version) using the following multiple choice question.
  To which gender identity do the participant most identify?
  * Female
  * Male
  * Transgender Female
  * Transgender Male
  * Other
  * Prefer Not to Answer
Study Population: A cohort of consecutive ED patients aged 18 years or more, treated for an acute pain condition present for less than 2 weeks (usual acute pain definition),and discharged with an opioid prescription will be included.
  In accordance to our pragmatic approach, we will exclude only patients with current use of opioids or chronic pain medication for a pre-existing condition or disease (e.g., cancer), because opioid dosage and/or pain mechanisms differ in these circumstances.
Sampling Method: Non-Probability Sample
Enrollment: 2240 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Quantity of opioids consumed during the acute pain phase (2 weeks) following ED discharge for each pain condition | During 14 days
  This will allow us to define the quantity of opioids needed to manage acute pain while limiting the quantity of unused pills available for potential misuse.

SECONDARY OUTCOMES:
Quantity of opioids prescribed to ED-discharged patients treated for different acute pain conditions | Baseline
  From physicians' prescriptions
Quantity of opioids to sufficiently supply a given percentage of patients for each pain condition | During 14 days
  Patient's questionnaire after 2 weeks and 14-diary on opioids consumption.
Quantity of unused opioids | At day 14
  Patient's questionnaire after 2 weeks
Quantity of patients that filled (initial or other) opioid prescriptions | At day 14
  Patient's questionnaire after 2 weeks
Quantity of patients using of coanalgesics or other substances (alcohol, cannabis…) to manage pain | During 14 days
  Patient's questionnaire after 2 weeks
Qualitative evaluation of the participants' reasons for stopping opioid consumption | During 14 days
  Patient's questionnaire after 2 weeks
Incidence and type of medication side effects during the 2-week period | During 14 days
  Patient's questionnaire after 2 weeks
Quantity of patients who revisit health services to obtain new prescription | During 14 days
  Patient's questionnaire after 2 weeks
Quantitive validation of the patients' self-report opioid consumption | At day 14
  Comparison of self-report comsumption and in person pill count after 2 weeks
Group-based trajectory modeling to determine pain intensity trajectory for each pain condition during the acute phase | During 14 days
  After 2 weeks. Average pain intensity for each patient will be measured using a 0-10 numerical rating scale for each of the 14-day diary.
  Group-based trajectory modeling will then be used to identify groups of patients with similar pattern of pain evolution over time without assuming the existence of a specific trend or number of groups.
Evaluate the chronic pain prevalence at 3 months among study participants assessed if certain profiles of pain intensity evolution over the14-day after emergency department (ED) discharge are predictive of chronic pain 3 months later. | 3 months
  After 90 days. Chronic pain will be defined as a pain intensity score at 3-month of >=4 and with moderate or severe functional disability using the pain disability index score (>40).
Assessed if certain profiles of pain intensity evolution over the14-day after emergency department (ED) discharge are predictive of chronic pain 3 months later | 3 months
  Pain intensity trajectories after 14 days and chronic pain at 3 months. Average pain intensity for each patient will be measured using a 0-10 numerical rating scale for each of the 14-day diary.
  Group-based trajectory modeling will then be used to identify groups of patients with similar pattern of pain evolution over time without assuming the existence of a specific trend or number of groups.
  Chronic pain will be defined as a pain intensity score at 3-month of >=4 and with moderate or severe functional disability using the pain disability index score (>40).

OTHER OUTCOMES:
Qualitative evaluation of participant's opioids storage and disposal | At day 14
  Patient's questionnaire after 2 weeks
Evaluate the participants' perception of opioid analgesia (patient, physician, nurse, and pharmacist) with a likert scale type survey | Baseline
  Survey with Likert style questions administered before start of recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Daoust, MD MSc, Principal Investigator — Université de Montréal
Locations (6):
- Canada (6):
  - Kingston General Hospital, Kingston, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Hôpital régional de Saint-Jérôme, Saint-Jérôme, Quebec
  - Hôpital de l'Enfant-Jésus, Québec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Daoust R, Paquet J, Perry JJ, Yan JW, Williamson D, Castonguay V, Lavigne G, Rouleau D, Lessard J, Cournoyer A; OPUM research group. How Does Self-Declared Chronic Pain Compare to Other Definitions? A Prospective Multicenter Study. Pain Res Manag. 2025 Jun 19;2025:5556400. doi: 10.1155/prm/5556400. eCollection 2025. PMID 40575042
- [Derived] Daoust R, Paquet J, Emond M, Iseppon M, Williamson D, Yan JW, Perry JJ, Huard V, Lavigne G, Lee J, Lessard J, Lang E, Cournoyer A; Quantity of Opioids for Acute Pain and Limit Unused Medication (OPUM) group on behalf of the Network of Canadian Emergency Researchers. Opioid prescribing requirements to minimize unused medications after an emergency department visit for acute pain: a prospective cohort study. CMAJ. 2024 Jul 14;196(25):E866-E874. doi: 10.1503/cmaj.231640. PMID 39009368
- [Derived] Daoust R, Paquet J, Williamson D, Perry JJ, Iseppon M, Castonguay V, Morris J, Cournoyer A. Accuracy of a self-report prescription opioid use diary for patients discharge from the emergency department with acute pain: a multicentre prospective cohort study. BMJ Open. 2022 Oct 28;12(10):e062984. doi: 10.1136/bmjopen-2022-062984. PMID 36307159